CLINICAL TRIAL: NCT03883880
Title: Salivary Interactions With Chemosensations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID (completed first intervention type only)
Sponsor: Purdue University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Cordelia Running, PhD, Assistant Prof. Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 082-011
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Diet, Food Choice, Taste
Keywords: diet; food choice; taste
MeSH Terms: interventions — epigallocatechin gallate; Linoleic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epigallocatechin gallate (Experimental): Epigallocatechin gallate solutions will be provided to participants to rinse with daily for two weeks. A control solution will be provided for two weeks as well. Order will be counterbalanced across participants and groups.
  Interventions: Other: Epigallocatechin gallate; Other: Epigallocatechin gallate control
- Linoleic acid (Experimental): Linoleic acid emulsion will be provided to participants to rinse with daily for two weeks. A control solution will be provided for two weeks as well. Order will be counterbalanced across participants and groups.
  Interventions: Other: Linoleic acid; Other: Linoleic acid control
- Capsaicin (Experimental): Capsaicin solutions will be provided to participants to rinse with daily for two weeks. A control solution will be provided for two weeks as well. Order will be counterbalanced across participants and groups.
  Interventions: Other: Capsaicin solution; Other: Capsaicin control

INTERVENTIONS:
Other: Epigallocatechin gallate — Colored solution prepared with epigallocatechin gallate to be consumed daily for two weeks during the epigallocatechin gallate intervention.
  Arms: Epigallocatechin gallate
Other: Epigallocatechin gallate control — Colored control solution to be consumed daily for two weeks during the epigallocatechin gallate intervention.
  Arms: Epigallocatechin gallate
Other: Linoleic acid — Colored emulsion prepared with linoleic acid to be consumed daily for two weeks during the linoleic acid intervention.
  Arms: Linoleic acid
Other: Linoleic acid control — Colored control solution to be consumed daily for two weeks during the linoleic acid intervention.
  Arms: Linoleic acid
Other: Capsaicin solution — Colored solution prepared with capsaicin to be consumed daily for two weeks during the capsaicin intervention.
  Arms: Capsaicin
Other: Capsaicin control — Colored control solution to be consumed daily for two weeks during the capsaicin intervention.
  Arms: Capsaicin

SUMMARY:
A counterbalanced, crossover design will be used to evaluate whether exposure to flavors vs. a control over time alters the perception of the flavor by changing an individual's salivary protein profile. Participants will complete 3 acute tasting protocols (baseline, after intervention 1, after intervention 2). The interventions will be with the flavor (epigallocatechin gallate, linolenic acid, capsaicin) or a control, in counterbalanced order, and will involve swishing and swallowing a solution of that sample 5 times per day for two weeks. Each of these flavors will be a separate sub-study.

DETAILED DESCRIPTION:
This study is designed to test the relationship between salivary proteins, flavor sensation, and flavor exposure. For this study, we will test the bitterness/astringency of epigallocatechin gallate (EGCG, a polyphenol), the oleogustus (fatty acid taste) of linolenic acid, and the spiciness of capsaicin in conjunction with the concentration of specific salivary proteins (initially: salivary proline rich proteins for EGCG intervention, lipocalin-1 for the other two, but other proteins may be identified in the post-hoc analysis of the salivary proteome). We will test whether higher expression of these specific salivary proteins correlates with lower intensity of these flavors. We will further attempt to confirm the role of these salivary proteins using food-sourced functional analogs for these proteins. We would expect the food-sourced protein to have the same effect on flavor as the salivary protein if our hypotheses about salivary proteins' influence on flavor are correct. Finally, we will also use denatured versions of the food-sourced proteins to again confirm that effects are due to the function of these proteins binding the flavor.

Additionally, we will repeatedly expose individuals to the flavors by having them rinse and swallow solutions of the flavor compounds multiple times per day for two weeks. We will then re-evaluate the sensory ratings and salivary protein profiles. Two weeks of rinsing and swallowing a control solution will be used as a control during this intervention (for each of the flavors of interest).

To collect saliva and establish bitterness/astringency perception, we will use an acute tasting protocol. Participants will rinse with water, then taste and swallow, then taste and expectorate a solution of the flavor of interest. Saliva will be frozen for later proteomic analysis. Next participants will taste solutions of: flavor, flavor with food analog, the flavor with denatured food analog, water, water with the food analog, and water with denatured food analog. The participants will rank these solutions in order from least intense to most intense for the flavor quality of interest (bitterness/astringency for EGCG). After this, participants will taste all 6 samples again, and rate each individually for the intensity of the bitterness/astringency. After a short wait, this tasting and intensity rating will be repeated. All tastings will be done in counterbalanced order, and solutions will be labeled with randomized 3-digit codes.

This acute tasting protocol will be done: at baseline, after 2 weeks on one intervention (repeated tasting of flavor or control), after 2 weeks on the other intervention.

ELIGIBILITY:
Inclusion Criteria:

* Agree to maintain current diet throughout intervention
* Agree to inform us if medication use changes during study.
* Willing and able to taste and consume samples, as well as take pictures to document use of the flavor during intervention.

Exclusion Criteria:

* Known issues with salivation, taste, or smell
* Taking medications other than birth control
* User of tobacco products or electronic cigarettes within the last 30 days

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Salivary proteins | 9 months per sub-study (intervention type)
  Subjects saliva will be collected at baseline, after the flavor intervention, and after control intervention (two weeks each, order counterbalanced) for each type of intervention (epigallocatechin gallate, linoleic acid, capsaicin). The proteomic composition of the saliva samples will be established, and used to evaluate relationships with other outcome measures.
Flavor intensity ratings | 9 months per sub-study (intervention type)
  Flavor intensities for the flavor of interest (bitterness/astringency, oleogustus, and spiciness) will be collected at baseline, after the flavor intervention, and after control intervention (two weeks each, order counterbalanced) for each type of intervention (epigallocatechin gallate, linoleic acid, capsaicin). Subjects will rate (in duplicate) the intensity of flavor from the following solutions: flavor in water, flavor in water with food-sourced salivary protein analog, flavor in water with denatured food-sourced salivary protein analog, water, water with food-sourced salivary protein analog , water with denatured food-sourced salivary protein analog. These ratings will be evaluated in context of the timeline of the exposure as well as the salivary proteome.
Flavor rankings | 9 months per sub-study (intervention type)
  Flavor rankings for the flavor of interest (bitterness/astringency, oleogustus, and spiciness) will be collected at baseline, after the flavor intervention, and after control intervention (two weeks each, order counterbalanced) for each type of intervention (epigallocatechin gallate, linoleic acid, capsaicin). Subjects will rank the following solutions from most to least intense: Flavor in water, flavor in water with food-sourced salivary protein analog, flavor in water with denatured food-sourced salivary protein analog, water, water with food-sourced salivary protein analog , water with denatured food-sourced salivary protein analog. These ranking data will be used an another method to gather information on what solutions are most intense to the subject, as the intensity ratings may have complications due to order effects during tastings. These rankings will also be evaluated in context of the timeline of the exposure as well as the salivary proteome.

CONTACTS AND LOCATIONS:
Overall Officials: Cordelia Running, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Davis LA, Running CA. Repeated exposure to epigallocatechin gallate solution or water alters bitterness intensity and salivary protein profile. Physiol Behav. 2021 Dec 1;242:113624. doi: 10.1016/j.physbeh.2021.113624. Epub 2021 Oct 14. PMID 34655570